CLINICAL TRIAL: NCT05804487
Title: ABL90 FLEX PLUS Clinical Precision Study for 15 Parameters in Adult Whole Blood
Status: Completed | Type: Observational
Sponsor: Radiometer Medical ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: DC-084059
Record Dates: First submitted 2023-03-26; First posted 2023-04-07 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2022-12

CONDITIONS: Diagnostic Test
Keywords: Blood gas

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples are collected to measure the pH, pCO2, pO2, cCa2+, cCl-, cK+, cNa+, cGlu, cLac, ctHb, sO2, FO2Hb, FMetHb, FCOHb and FHHb parameters in adult whole blood.
  Samples are destroyed when measurements are completed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: ABL90 FLEX PLUS analyser running SW3.5 MR2. — The ABL90 FLEX PLUS analyzer is a portable, automated analyzer that measures pH, blood gases, electrolytes, metabolites, and oximetry in whole blood - utilizing 3 measuring modes (syringe, short probe, and capillary mode) to measure samples from a syringe, test tube or a capillary tube. The analyzer provides results for 17 parameters in 35 seconds using 65 μL heparinized whole blood.

SUMMARY:
Conducting the ABL90 FLEX PLUS Clinical Precision Study for 15 Parameters in Adult Whole Blood is to validate performance claims for precision in heparinized whole blood for 15 parameters: pH, pCO2, pO2, cCa2+, cCl-, cK+, cNa+, cGlu, cLac, ctHb, sO2, FO2Hb, FMetHb, FCOHb, and FHHb, while being influenced by testing environment that is representative of intended use environment, site variability, and operator variability in a point-of-care (POC) setting.

The investigational device is the ABL90 FLEX PLUS (Figure 1) incl. consumables, running SW3.5 MR2, manufactured by Radiometer Medical ApS The study is being conducted in Denmark and in total, a minimum of 105 subjects are to be enrolled to provide successful measurement values from 3 different sites.

DETAILED DESCRIPTION:
The conduct of the clinical study is to determine repeatability of each parameter using replicate measurements from heparinized whole blood samples measured by intended users in syringe, short probe, and capillary modes available for ABL90 FLEX PLUS, in a POC setting.

The study endpoint is repeatability (SD) in whole blood for each parameter, measuring mode and parameter level, pooled across sites. Participating sites are intensive care wards, and the adult patients (≥18 years old ) are admitted to the hospital with low (moderate hypo), normal, or elevated (moderate hyper) concentrations of the 15 parameters covering the reportable range as much as possible. For collecting whole blood samples, the subject is required to have either arterial or Central Venus Catheter (CVK) lines established as part of standard of care to minimize the risk to the patient.

Each sample of 1.5 mL whole blood is used to complete 2 replicates per run (Each sample will be measured twice on the selected mode during 1 run). Samples to be measured in syringe mode are measured from a syringe, or samples to be measured in capillary mode are transferred to capillary tubes from a syringe and measured from a capillary tube.

Part 1:

1. Samples collected from 20 subjects (patients).
2. 6 samples of whole blood are collected from each subject (3 samples for Run 1 and 3 samples for Run 2).
3. Minimum 40 whole blood samples to be measured in S65 syringe mode (20 subjects x 2 samples per subject).
4. Minimum 40 whole blood samples to be measured in SP65 short-probe mode (20 subjects x 2 samples per subject).
5. Minimum 40 whole blood samples to be measured in C65 capillary mode (20 subjects x 2 samples per subject).
6. Minimum 120 whole blood samples to be measured in all 3 modes free of errors. If errors occur, a new sample needs to be collected.

Part 2:

1. Samples collected from 15 subjects (patients or donate blood).
2. 9 samples of whole blood are collected from each subject. (3 samples in S65 mode, 3 samples in SP65 mode, 3 samples transferred into 6 capillary tubes in C65 mode).
3. Minimum 45 whole blood samples to be measured in S65 syringe mode (15 subjects x 3 samples per subject).
4. Minimum 45 whole blood samples to be measured in SP65 short-probe mode (15 subjects x 3 samples per subject).
5. Minimum 45 whole blood samples to be measured in C65 capillary (15 subjects x 3 samples per subject).
6. Minimum 135 whole blood samples to be measured in all 3 modes free of errors. If errors occur, a new sample needs to be collected.

Minimum 255 (heparinized) whole blood samples obtained from adult patients or donate blood are required for this study from each site.

This study will evaluate 2-3 levels per parameter covering the moderate hypo, normal and moderate hyper range.

Three POC users, such as a nurse, a physician, or a therapist perform the measurements in an equal range.

Samples are collected to measure the pH, pCO2, pO2, cCa2+, cCl-, cK+, cNa+, cGlu, cLac, ctHb, sO2, FO2Hb, FMetHb, FCOHb, and FHHb parameters in heparinized whole blood. Samples are destroyed when measurements are completed.

The ABL90 FLEX PLUS analyzer is a portable, automated analyzer that measures pH, blood gases, electrolytes, metabolites, and oximetry in whole blood - utilizing 3 measuring modes (syringe, short probe, and capillary mode) to measure samples from a syringe, test tube or a capillary tube. The analyzer provides results for 17 parameters in 35 seconds using 65 μL heparinized whole blood.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older.
* Obtained informed consent from subject or from relative(s) able to understand information given and willing and able to voluntary give their consent to participate in this study.
* Subject shall have an arterial or a CVK line established as a part of the standard care.
* Subject evaluated as suitable according to the protocol and for the study by the principal investigator or designee.

Exclusion Criteria:

* Subjects where sample collection is evaluated by principal investigator or designee to impose an unnecessary risk.
* Subjects, who are pregnant or breastfeeding.
* Subjects who have been previously enrolled into this study.
* Subjects taking medications listed in Appendix 1 within 72 hours of the sample collection
* Subjects with known infectious disease such as Hepatitis C or HIV (to ensure the operator safety)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old ) admitted to the hospital with low (moderate hypo), normal, or elevated (moderate hyper) concentrations of the 15 parameters covering the reportable range as much as possible.
  For collecting whole blood samples, the subject is required to have either arterial or Central Venus Catheter (CVK) lines established as part of standard of care to minimize the risk to the patient.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Repeatability (SD) in whole blood for each parameter, measuring mode and parameter level, pooled across sites. | 4 - 6 hours
  Repeatability of each parameter (pH, pCO2, pO2, cCa2+, cCl-, cK+, cNa+, cGlu, cLac, ctHb, sO2, FO2Hb, FMetHb, FCOHb and FHHb) using replicate measurements from heparinized whole blood samples measured by intended users in syringe, short probe, and capillary modes available for ABL90 FLEX PLUS, in a POC setting.

CONTACTS AND LOCATIONS:
Overall Officials: Tejs Jansen, Principal Investigator — External Coordinating Principal Investigator
Locations (1):
- Tejs Jansen, Copenhagen, Østerbro, Denmark

IPD SHARING:
Plan to Share IPD: Yes
When the Clinical Study Report has been finalized, Data result will be available for public on platforms and in articles.
Supporting Information: CSR
Time Frame: The data will become available within a year after end of study.